CLINICAL TRIAL: NCT00824603
Title: Impact of CME Program on Self-Reported Confidence and Use of Insulin in Persons With Type 2 Diabetes
Brief Title: Impact of Continuing Medical Education (CME) Insulin Program
Status: Completed | Type: Observational
Sponsor: HealthPartners Institute (Other)
Collaborators: International Diabetes Center at Park Nicollet (Other); Eli Lilly and Company (Industry); Novo Nordisk A/S (Industry); United Health Care (Unknown); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 03425-06-C
Record Dates: First submitted 2009-01-15; First posted 2009-01-19 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2013-08

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- primary care provider: attending insulin CME Training

SUMMARY:
The purpose of this study is to determine if a continuing medical education (CME) program can change primary care providers' use of insulin therapy - their confidence in selecting doses and engagement of patients in the decision making as to whether to initiate insulin therapy.

DETAILED DESCRIPTION:
We will determine whether attendees' self-reported confidence and use of insulin with persons with type 2 diabetes changes after they attend the CME program. Specifically, we will address the following questions:

Question 1. Clinical guidelines. Is insulin initiated earlier (at a lower A1C)?

Question 2. Decision-making. Does confidence in selecting a starting insulin regimen change? Does confidence in selecting a starting insulin dose change? Does confidence in adjusting insulin change? Does confidence in discussion nutrition guidelines change?

Question 3. Application. Do more patients start using insulin? Who usually selects starting dose? How is starting dose selected? How often is insulin adjusted?

Question 4. Resources. How available are protocols for insulin use? How available is adequate time to monitor insulin therapy? How available is staff to teach insulin injections? How available is staff to help adjust insulin?

ELIGIBILITY:
Inclusion Criteria:

* primary care provider attending CME training

Exclusion Criteria:

-

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care providers affiliated with the participating healthcare organizations were invited to attend.
Sampling Method: Non-Probability Sample
Enrollment: 294 (Actual)
Dates: Start 2006-06; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
We will determine whether attendees' self-reported confidence and use of insulin with persons with type 2 diabetes changes after they attend the CME program. | pre program survey & 2-4 month post program survey

SECONDARY OUTCOMES:
pre-CME training level of patient's A1c when starting insulin therapy compared to post-CME training level of patient's A1c when starting insulin therapy | pre program survey and 2-4 month post program survey

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Powers, PhD, Principal Investigator — International Diabetes Center at Park Nicollet
Locations (1):
- International Diabetes Center, Minneapolis, Minnesota, United States